CLINICAL TRIAL: NCT06111807
Title: GUIding Multi-moDal thErapies Against MRD by LiquidBiopsies in Non Small Cell Lung Cancer- GUIDE.MRD-03-NSCLC
Brief Title: Clinical Validation and Benchmarking of Top Performing ctDNA Diagnostics - Stage III NSCLC
Acronym: MRD-LUNG
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: LungenClinic Grosshansdorf (Other); Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: GUIDE.MRD-03-NSCLC
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer Stage III
Keywords: Circulating tumor DNA; ctDNA diagnostics; Minimal residual disease; Sensitivity; Specificity; complete pathological response
MeSH Terms: conditions — Lung Neoplasms; Neoplasm, Residual; Hypersensitivity; Pathologic Complete Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Full blood samples processed into plasma, buffy coat,and serum Formalin-fixed paraffin-embedded tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Chemo-radiotherapy: Stage 3 NSCLC eligible for chemoradiotherapy
  Interventions: Diagnostic Test: ctDNA
- Neoadjuvant and surgery: Stage 3 NSCLC eligible for neoadjuvant chemo-immunotherapy followed by surgery
  Interventions: Diagnostic Test: ctDNA
- Surgery and adjuvant immunotherapy: Stage 3 NSCLC eligible for surgery followed by immunotherapy
  Interventions: Diagnostic Test: ctDNA

INTERVENTIONS:
Diagnostic Test: ctDNA — ctDNA will be tested retrospectively, no treatment decisions will be made prospectively

SUMMARY:
Improving personalized cancer treatments and finding the best strategies to treat each patient relies on using new diagnostic technologies. Currently, for non small cell lung cancer (NSCLC), the methods used to decide who gets additional post radical (surgery or definite chemo-radiotherapy) treatment are suboptimal. Some patients get too much treatment, while others do not get enough.

There is a new way to explore if there is any cancer left in a patient's body using circulating tumor DNA (ctDNA) detected in blood samples. This can help decide who needs more treatment. Even though many tests have been developed, it has yet to be determined which test performs best at relevant time points.

The GUIDE.MRD consortium is a group of experts, including scientists, technology, and pharmaceutical companies. The consortium is working on creating a reliable standard for the ctDNA tests, validating their clinical utility, and collecting data to help decide on the best treatment for each patient.

GUIDE.MRD-03-NSCLC is a part of the GUIDE.MRD project.

DETAILED DESCRIPTION:
GUIDE.MRD-03-NSCLC is a part of WP3 of the overarching GUIDE.MRD project. Each study chair has a local clinical trial protocol where patients are recruited. After the end of recruitment, samples will be analyzed under the GUIDE.MRD consortium.

The overall aim of GUIDE.MRD is to investigate the clinical utility of ctDNA analysis to predict and guide the choice of multi-modal therapies prospectively. The fundamental steps towards this aim are assessment and benchmarking of the many available ctDNA diagnostics to identify the best-suited tests for clinical application. Clinical samples will be used to benchmark ctDNA diagnostics and assess their true clinical performance. The samples should reflect clinical situations where the ctDNA diagnostics are particularly useful, such as post-operatively, post-adjuvant, during chemotherapy, and longitudinally during post-treatment surveillance. In these situations, ctDNA diagnostics could be used to either monitor treatment response (in case of MRD after surgery or definite chemoradiotherapy) or to identify relapse at an early time point. Based on ctDNA information, medical treatment could be changed, or radiology could be used to reveal the location of residual disease.

The rationale for the observational clinical study GUIDE.MRD-03-NSCLC is to prospectively collect the clinical samples needed to enable assessment of the performance of ctDNA diagnostics in the setting of non small cell lung cancer (NSCLC). There are three main scenarios where ctDNA diagnostic is useful in NSCLC in a MRD setting:

For this study stage III NSCLC will be included treated with curative intent using:

1. chemo-radiotherapy (concurrent or sequential) followed by adjuvant immunotherapy. This patient group is particularly relevant because adjuvant therapy is recommended for all stage III patients (in some countries for those with PD-L1>1% only), due to their high recurrence risk around 58%. Additionally, most of these do not need therapy at all, because they were already cured by chemo-radiotherapy alone, which leads to substantial overtreatment. Furthermore, the 58% of patients who recur despite both chemoradiotherapy and adjuvant immunotherapy, probably could benefit from further multimodal therapies. The challenge is, however, that currently there is no marker in clinical use that can identify those patients with residual disease and need for therapy. Circulating tumor DNA is potentially such a marker.
2. Neoadjuvant treatment followed by surgery (or radiotherapy with curative intent). In this setting up to 30% have a complete pathological response (pCR). These patients are probably cured by the neoadjuvant treatment alone, where surgery thus might have been avoided if the MRD biomarker would be sensitive enough. Patients that did not receive a pCR do worse with a median overall survival around 24 month even when they are treated with immunecheckpoint inhibitors adjuvantly. Better strategies for selecting patients and treatments are urgently needed here as well. Again ctDNA could be a marker that may help here when sensitive enough to select those that are negative for no adjuvant and those that are positive for ctDNA guided multimodality treatment.
3. Surgery followed by adjuvant chemotherapy and immunotherapy. Patients in this setting may be treated by immunotherapy adjuvantly only when PD-L1>1% (FDA) or PD-L1>50% (EMA). Also here recurrence risk is high around 50%. Additionally, most of these do not need therapy at all, because they were already cured by surgery alone, which leads to substantial overtreatment. Furthermore, the 50% of patients who recur despite both surgery and adjuvant therapy, probably could benefit from further multimodal therapies. The challenge is, however, that currently there is no marker in clinical use that can identify those patients with residual disease and need for therapy. Circulating tumor DNA is potentially such a marker.

However, currently, it is unknown, which, if any,of the many different ctDNA diagnostics developed in recent years have the required, performance to provide clinical utility in the management in these settings of stage III NSCLC.

Primary objectives:

To assess the performance of ctDNA diagnostics using samples collected at four to five -landmark time-points "baseline"; "post neoadjuvant treatment"; "post-surgery or chemoradiotherapy"; "post-adjuvant therapy" and "at the end of study or disease progression".Sensitivity, specificity, and positive and negative predictive values of the ctDNA diagnostics will be determined to enable a head-to-head performance assessment and benchmarking of ctDNA diagnostics.

Secondary objectives To assess the ctDNA stratified 3-year recurrence-free survival (RFS). To assess the lead time between ctDNA detection and clinical recurrence. To assess the capacity of the ctDNA diagnostics to predict response to neoadjuvant therapy.

To assess the capacity of the ctDNA diagnostics to predict response to adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC, clinical tumor stage III (cT1-4, cN0-3, M0).
* Patient 18 years or older.
* Scheduled for curative intent treatment (surgery and/or radiotherapy).
* Patient able to understand and sign written informed consent.
* Baseline contrast enhanced CT thorax abdomen (or PET/CT), MRI (or CT) brain, Pulmonary function tests (at least FEV1 and DLCO/KCO).
* Ability to obtain sufficient tumor material (≥50ng tumor DNA, FFPE ). Either at baseline or after surgery.

Exclusion Criteria:

* Verified distant metastases.
* With synchronous NSCLC cancer and non-NSCLC cancer (except skin cancer other than melanoma).
* With other cancers (excluding NSCLC or skin cancer other than melanoma, or cancers treated curatively with follow up of more than 5 years without recurrence).
* Patients who are unlikely to comply with the protocol (e.g. uncooperative attitude), inability to return for subsequent visits) and/or otherwise considered by the Investigator to be unlikely to complete the study.
* No tissue sample available for the project, or tumor content in the tissue sample is <20%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage III NSCLC with curative intent treatment
Sampling Method: Non-Probability Sample
Enrollment: 248 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Collection of clinical plasma samples at relevant time points | 8 months after end of recruitment
  For head-to-head performance assessment and benchmarking of ctDNA diagnostics

SECONDARY OUTCOMES:
The 3-year recurrence-free survival | 3 years after end of recruitment
  recurrence free survival by RECIST1.1
Lead time between ctDNA detection and clinical recurrence | 3 years after end of recruitment
  recurrence by RECIST1.1
Prognostic value of ctDNA analysis at relevant time points | 3 years after end of recruitment
  for complete pathological response, disease progression, event free and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Abdo, MD, Study Chair — LungenClinic Grosshansdorf; Paul Hofman, MD, PhD, Study Chair — Centre Hospitalier Universitaire (CHU) de Nice
Locations (6):
- France (2):
  - Centre Hospitalier Universitaire de Nice, Nice, Nice
  - Antoine Lacassagne Center, Nice, Nice
- Department of thoracic oncology- LungenClinic Großhansdorf, Großhansdorf, Grosshansdorf, Germany
- Netherlands (3):
  - Isala, Zwolle, Overijssel
  - University Medical Center Groningen, Departments of Pulmonology and Pathology, Groningen, Provincie Groningen
  - Ommelander Ziekenhuis Groningen, Scheemda, Provincie Groningen

IPD SHARING:
Plan to Share IPD: Undecided
will be anonymized

REFERENCES:
- See also: Webpage of the GUIDE.MRD project — http://www.guidemrd-horizon.eu/